CLINICAL TRIAL: NCT06909240
Title: Progressive Gait Training After First-time Deep Venous Thrombosis: Clinical Effectiveness and Involved Mecanisms (The DVT-Cph RCT)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hvidovre University Hospital (Other)
Responsible Party: Principal Investigator, Ove Andersen, Professor, Hvidovre University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H-22017283 / 2.3
Record Dates: First submitted 2025-03-27; First posted 2025-04-03 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Deep Vein Thrombosis (DVT)
Keywords: Physical activity
MeSH Terms: conditions — Venous Thrombosis; Motor Activity | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental)
  Interventions: Other: Progressive gait training
- Control (Active Comparator)
  Interventions: Other: Standard Care (in control arm)

INTERVENTIONS:
Other: Progressive gait training — The focus of the intervention is on exercises that can improve venous return, and consists of progressive gait training at moderate and high intensity as well as guidance on progressive gait training. The training program is inspired by the WHO's recommendations for physical activity. The training program consists of a 14-day introductory period based on an initial interview with a physiotherapist, where the aim is to obtain 30 mins/day of gait training at moderate intensity. After 14 days, the patient receives physiotherapist guidance via telephone on progressive gait training and is introduced to the next period of 14 days, where the activity level is maintained, and the goal is to further achive 2 x 20 mins/week of muscle-strengtening activities at moderate or greater intensity. After one and two months of training, the patient will be guided via telephone on maintaining their current level of physical activity or possibly on further progression.
  Arms: Intervention
Other: Standard Care (in control arm) — Standard care encompasses standard diagnostics with compression ultrasound examination, and a treatment procedure with anticoagulant medication, and compression stockings class III. Standard care also involves visits to the outpatient anticoagulation clinic, where patients with DVT are required to attend treatment sessions within the first 14 days and 90 days after diagnosis. Standard care will serve as a comparator to reflect the current treatment regimen.
  Arms: Control

SUMMARY:
The DVT-Cph RCT aims to investigate:

1. if progressive gait training in combination with standard care is superior to standard care on quality of life in patients with first time lower extremity deep venous thrombosis (clinical effectiveness part).
2. the association between progressive gait training and disease progression, late complications such as post throbotic syndrome, and severity of venous thromboembolism conditions in patients with first time lower extremity deep venous thrombosis (mechanistic part).

DETAILED DESCRIPTION:
The DVT-Cph RCT will be qualified by a preceeding feasibility trial (NCT05761119) that aims to investigate: (1) the feasibility of the intervention and trial procedures using quantitative outcomes, and (2) patient experiences with and attititudes towards the intervention using qualitative interviews.

Simultaneously with the RCT, a prospective cohort study (The DVT-Cph cohort study; NCT05789108) will investigate and characterize acutely admitted patients with deep venous thrombosis via inflammatory, anti-inflammatory, immunological and ageing biomarkers to gain a better understanding of options about prevention and treatment of long-term complications. Patients enrolled in the feasibility trial as well as in the DVT-Cph RCT can also enroll in the DVT-Cph cohort study to utilize study synergy and enhance research information gain.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or above
* First time lower extremity DVT
* Hospitalized at the Emergency Department
* Can cooperate cognitively and physically (patient reported)

Exclusion Criteria:

* Patients without a Danish social security number
* Terminal patients
* Patients who do not understand or speak Danish

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Estimated)
Dates: Start 2025-11-15 (Actual); Primary Completion 2028-04-01 (Estimated); Study Completion 2030-02-01 (Estimated)

PRIMARY OUTCOMES:
The Venous Insufficiency Epidemiological and Economic Study - Quality of Life/Symptoms (VEINES-QOL/Sym) questionnaire | Change from baseline to 3 months after discharge (end of intervention)
  The VEINES-Qol is a validated disease-specific questionnaire for measuring quality of life among patients with a venous disease (Lamping D et al., 2003).

SECONDARY OUTCOMES:
The Venous Insufficiency Epidemiological and Economic Study - Quality of Life/Symptoms (VEINES-QOL/Sym) questionnaire | Change from baseline to 12 and 24 months after discharge
  The VEINES-Qol is a validated disease-specific questionnaire for measuring quality of life among patients with a venous disease (Lamping D et al., 2003).
Health status measured by the EuroQol instrument (EQ-5D-5L) | Change from baseline to 3 (end of intervention), 12, and 24 months after discharge
  The EuroQol-5D-5L consists of five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression, along with a visual analog scale (EuroQol-VAS). Each dimension includes five response levels, ranging from no problems to extreme problems. The responses are converted into an index value that reflects the individual's health status in comparison to the general population (norm data)(EuroQol Group, 1990; Herdman M et al., 2011 ). EuroQol-VAS measures health on a scale from 0 (worst imaginable health) to 100 (best imaginable health).
Pain measured by the Visual Analogue Scale | Recurrent weekly outcome from baseline to 3 months after discharge (end of intervention)
  Pain measured by the VAS ranging from "no pain" (score of 0) to "worst imaginable pain" (score of 10). VAS scores are reported weekly by questionnaires sent by email or text message during the intervention as well as during follow up visits. Patients are asked to mark a point on the scale that represents their perception of the pain that they are feeling. Three different variables are collected: I) Current pain, II) lowest perceived pain within the last week and III) highest perceived pain within the last week
Oedema | Change from baseline to 3 (end of intervention), 12, and 24 months after discharge
  Oedema on the symptomatic side compared to the healthy side. Oedema is measured by a medical doctor at the calf 10 cm below the tibial tuberosity on both legs
Development of Post Thrombotic Syndrome (PTS) measured by the Villalta-score | Change from baseline to 3 (end of intervention), 12, and 24 months after discharge (end of intervention)
  The Villalta-score consists of five patient-related venous symptoms and six clinician-rated physical signs. Each of the 11 items is graded on a scale from 0 (not present) to 3 points (severe) rendering a maximum total score of 33 points (Lee A et.al., 2021). The points are summed and results in a total score. Subject are classified as having developed PTS if the score is ≥ 5 points or if a venous ulcer is present, in the leg ipsilateral to the initial DVT at a single assessment (Kahn SR et al., 2014, Kahn SR et al., 2009) , either at 90 days (+/-30 days), 12 months (+/- 30 days) or 24 months (+/- 30 days) at the follow-up visits. The severity of PTS can further be categorized as mild (Villalta score 5-9), moderate (score between 10-14), or severe PTS/venous ulcer (score ≥ 15).
Number of DVT related hospital contacts | From baseline to 3, 12, and 24 months after discharge

OTHER OUTCOMES:
Chronic inflammation | Change from baseline to 3, 12, and 24 months after discharge
  Chronic inflammation will be measured based on the soluble urokinase Plasminogen Activator Receptor (suPAR). suPar will be measured using standard immunoassays. Plasma levels of inflammation biomarkers and anti-inflammation biomarkers will be analysed at Department of Clinical Research, Acute CAG, Copenhagen University Hospital Amager and Hvidovre

CONTACTS AND LOCATIONS:
Overall Officials: Helle Juul-Larsen, Ph.D., Principal Investigator — Hvidovre University Hospital; Mette Merete Pedersen, Ph.D., Principal Investigator — Hvidovre University Hospital; Izzet Altinas, M.D., Principal Investigator — Hvidovre University Hospital
Locations (1):
- Hvidovre University Hospital, Hvidovre, Capital Region, Denmark

IPD SHARING:
Plan to Share IPD: No
Public deposition of raw data points is not possible due to Denmarks national legislation (Data Protection Act § 10 and Data Disclosure Proclamation Act) which outline that we can only transfer pseudonymized data to the Journal after the Data Protection Authorities approval (Data Protection Act § 10, section 3, nr. 3.).
  Reviewers and others may obtain access to the data by request, and after the Danish Data Protection Agency has approved of the data transfer from the Capital Region to the Journal. If others are to gain access to the pseudonymized data, the Journal shall ensure that is an adequate legal basis to share the Capital Regions data and ensure that the data is only being processed for scientific research purposes.

REFERENCES:
- [Background] EuroQol Group. EuroQol--a new facility for the measurement of health-related quality of life. Health Policy. 1990 Dec;16(3):199-208. doi: 10.1016/0168-8510(90)90421-9. PMID 10109801
- [Background] Kahn SR. Measurement properties of the Villalta scale to define and classify the severity of the post-thrombotic syndrome. J Thromb Haemost. 2009 May;7(5):884-8. doi: 10.1111/j.1538-7836.2009.03339.x. Epub 2009 Mar 6. PMID 19320818
- [Background] Kahn SR, Comerota AJ, Cushman M, Evans NS, Ginsberg JS, Goldenberg NA, Gupta DK, Prandoni P, Vedantham S, Walsh ME, Weitz JI; American Heart Association Council on Peripheral Vascular Disease, Council on Clinical Cardiology, and Council on Cardiovascular and Stroke Nursing. The postthrombotic syndrome: evidence-based prevention, diagnosis, and treatment strategies: a scientific statement from the American Heart Association. Circulation. 2014 Oct 28;130(18):1636-61. doi: 10.1161/CIR.0000000000000130. Epub 2014 Sep 22. No abstract available. PMID 25246013
- [Background] Herdman M, Gudex C, Lloyd A, Janssen M, Kind P, Parkin D, Bonsel G, Badia X. Development and preliminary testing of the new five-level version of EQ-5D (EQ-5D-5L). Qual Life Res. 2011 Dec;20(10):1727-36. doi: 10.1007/s11136-011-9903-x. Epub 2011 Apr 9. PMID 21479777
- [Background] Lee A, Gu CS, Vedantham S, Kearon C, Blostein M, Kahn SR. Performance of two clinical scales to assess quality of life in patients with post-thrombotic syndrome. J Vasc Surg Venous Lymphat Disord. 2021 Sep;9(5):1257-1265.e2. doi: 10.1016/j.jvsv.2021.01.017. Epub 2021 Feb 4. PMID 33548557
- [Background] Lamping DL, Schroter S, Kurz X, Kahn SR, Abenhaim L. Evaluation of outcomes in chronic venous disorders of the leg: development of a scientifically rigorous, patient-reported measure of symptoms and quality of life. J Vasc Surg. 2003 Feb;37(2):410-9. doi: 10.1067/mva.2003.152. PMID 12563215